CLINICAL TRIAL: NCT01469429
Title: Food-Based Modulation of Biomarkers in Human Tissues at High-Risk for Oral Cancer
Brief Title: Phase 1b Food Based Modulation of Biomarkers in Human Tissues at High-Risk for Oral Cancer.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Amit Agrawal, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OSU-07085; NCI-2011-03226 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-10-27; First posted 2011-11-10 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Metastatic Squamous Neck Cancer With Occult Primary Squamous Cell Carcinoma; Salivary Gland Squamous Cell Carcinoma; Stage 0 Hypopharyngeal Cancer; Stage 0 Laryngeal Cancer; Stage 0 Lip and Oral Cavity Cancer; Stage 0 Nasopharyngeal Cancer; Stage 0 Oropharyngeal Cancer; Stage 0 Paranasal Sinus and Nasal Cavity Cancer; Stage I Salivary Gland Cancer; Stage I Squamous Cell Carcinoma of the Hypopharynx; Stage I Squamous Cell Carcinoma of the Larynx; Stage I Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage I Squamous Cell Carcinoma of the Nasopharynx; Stage I Squamous Cell Carcinoma of the Oropharynx; Stage I Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage I Verrucous Carcinoma of the Larynx; Stage I Verrucous Carcinoma of the Oral Cavity; Stage II Salivary Gland Cancer; Stage II Squamous Cell Carcinoma of the Hypopharynx; Stage II Squamous Cell Carcinoma of the Larynx; Stage II Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage II Squamous Cell Carcinoma of the Nasopharynx; Stage II Squamous Cell Carcinoma of the Oropharynx; Stage II Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage II Verrucous Carcinoma of the Larynx; Stage II Verrucous Carcinoma of the Oral Cavity; Stage III Salivary Gland Cancer; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Nasopharynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Verrucous Carcinoma of the Larynx; Stage III Verrucous Carcinoma of the Oral Cavity; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IVA Salivary Gland Cancer; Stage IVA Squamous Cell Carcinoma of the Larynx; Stage IVA Oral Cavity Squamous Cell Carcinoma; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Stage IVA Nasal Cavity and Paranasal Sinus Cancer; Stage IVA Verrucous Carcinoma of the Larynx; Stage IVA Verrucous Carcinoma of the Oral Cavity; Stage IVB Salivary Gland Cancer; Stage IVB Squamous Cell Carcinoma of the Larynx; Stage IVB Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Oropharynx; Stage IVB Oral Cavity Squamous Cell Carcinoma; Stage IVB Verrucous Carcinoma of the Larynx; Stage IVB Verrucous Carcinoma of the Oral Cavity; Stage IVC Salivary Gland Cancer; Stage IVC Squamous Cell Carcinoma of the Larynx; Stage IVC Oral Cavity Squamous Cell Carcinoma; Stage IVC Squamous Cell Carcinoma of the Oropharynx; Paranasal Sinus and Nasal Cavity Squamous Cell Carcinoma; Stage IVC Verrucous Carcinoma of the Larynx; Stage IVC Verrucous Carcinoma of the Oral Cavity; Tongue Cancer
Keywords: oral cancer
MeSH Terms: conditions — Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Paranasal Sinus Neoplasms; Tongue Neoplasms | interventions — Chemoprevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm I (Lozenge placebo) (Placebo Comparator): Patients receive lozenge placebo PO QID.
  Interventions: Other: placebo; Other: laboratory biomarker analysis; Other: questionnaire administration
- Arm II (LBR lozenge) (Experimental): Patients receive lyophilized black raspberries lozenge PO (8gms/day)
  Interventions: Other: laboratory biomarker analysis; Other: questionnaire administration; Drug: chemoprevention
- Arm III (Saliva Substitute placebo) (Placebo Comparator): Patients receive Saliva Substitute placebo PO QID.
  Interventions: Other: laboratory biomarker analysis; Other: questionnaire administration; Other: placebo
- Arm IV (LBR Saliva Substitute) (Experimental): Patients receive lyophilized black raspberries Saliva Substitute PO (8gms/day).
  Interventions: Other: laboratory biomarker analysis; Other: questionnaire administration; Drug: chemoprevention

INTERVENTIONS:
Other: placebo — Receive lozenge placebo PO
  Other Names: PLCB
  Arms: Arm I (Lozenge placebo)
Other: laboratory biomarker analysis — Correlative studies
Other: questionnaire administration — Ancillary studies
Drug: chemoprevention — Receive LBR lozenge PO
  Other Names: cancer chemoprevention; chemoprevention of cancer
  Arms: Arm II (LBR lozenge)
Drug: chemoprevention — Receive LBR Saliva Substitute PO
  Other Names: cancer chemoprevention; chemoprevention of cancer
  Arms: Arm IV (LBR Saliva Substitute)
Other: placebo — Receive Saliva Substitute placebo PO
  Other Names: PLCB
  Arms: Arm III (Saliva Substitute placebo)

SUMMARY:
This randomized phase I/II trial studies the side effects and best way to give lyophilized black raspberries in preventing oral cancer in high-risk patients previously diagnosed with stage I-IV or in situ head and neck cancer. Chemoprevention is the use of certain drugs to keep cancer from forming. The use of lyophilized black raspberries may prevent oral cancer. Studying samples of oral cavity scrapings, blood, urine, and saliva in the laboratory from patients receiving lyophilized black raspberries may help doctors learn more about changes that occur in DNA and the effect of lyophilized back raspberries on biomarkers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the adherence of post-surgical head and neck (HN) cancer patients to clinical trial design expectations and define tolerability and potential adverse effects of long-term black raspberry administration in this patient cohort.

II. Determine the effects of dose and delivery vehicle on the degree of uptake of black raspberry components in target oral tissues of post-surgical HN cancer patients over time and determine the relationships between adherence/exposure data and uptake.

III. Determine the ability of black raspberries to modulate patterns of gene expression within key regulatory pathways in "at-risk normal" oral mucosa of post-surgical HN cancer patients that would favor the inhibition, delay or reversal of oral carcinogenesis.

IV. Determine the persistence of modulation of "berry-responsive genes" for 2 years following commencement of black raspberry treatment and preliminarily define rate of recurrence and second primary oral cancers in a former oral cancer patient sub-cohort.

OUTLINE: Patients are randomized to 1 of 4 treatment arms.

ARM I: Patients receive lozenge placebo orally (PO) four times daily (QID).

ARM II: Patients receive lyophilized black raspberries lozenge PO QID.

ARM III: Patients receive Saliva Substitute placebo PO QID.

ARM IV: Patients receive lyophilized black raspberries Saliva Substitute PO QID.

In all arms, treatment continues for 6 months. Oral cavity scrapings, blood, urine, and saliva samples are collected periodically for laboratory analyses.

After completion of study treatment, some patients are followed up at weeks 1-5 and then at 2, 6, 12, and 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects includes all adult HN cancer patients who have been previously diagnosed with Stage 1-4 and in-situ squamous cell carcinoma within the past 36 months (mos); with or without further adjuvant therapy and have been determined to be disease free at the time of consent
* Patients must be able to take nutrition/medications orally
* Have no prior history of intolerance or allergy to berry or berry-containing products
* Patients taking cyclooxygenase (COX)-1/COX-2 inhibitors (Indomethacin, Ibuprofen, celebrex) chronically, herbal supplements, who cannot be taken off the medication/supplement due to their clinical condition are eligible to participate in the study but should document daily doses of these medications in their logbooks

Exclusion Criteria:

* History of intolerance (including hypersensitivity or allergy) to berry or berry-containing products
* Inability to take oral nutrition/liquids or history of aspiration pneumonia
* Pregnant women: Although there are no known adverse effects of black raspberries upon the fetus, if patients become pregnant during period of lyophilized black raspberries (LBR) administration, then LBR will be discontinued and patient will be removed from the study; we should however emphasize, given this is a food based-study, that risks are likely extremely low even though a participant should become pregnant; as such, we are not recommending active contraception for women, but rather if participants become pregnant, that they notify their study doctor, and that they will likely be removed from study; there are no expected or logical risks if men were to father a child, and as such, no contraception will be recommended for men
* Inability to grant informed consent
* Strict Vegetarians will be excluded from the study; it was found that consuming one portion per day of fruit or vegetables resulted in a significant decrease in oral cancer incidence; in those persons consuming multiple portions each day, there was a 50% reduction in risk; we assume that strict vegetarians will consume multiple portions each day of foods with chemopreventive activity and therefore inclusion of these individuals would have a negative impact on the study; there are several reports in the literature that herbal or multivitamin/mineral supplements have no effect on oral cancer incidence

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-09-04 (Actual); Primary Completion 2014-09-17 (Actual); Study Completion 2014-09-17 (Actual)

PRIMARY OUTCOMES:
Define tolerability and potential adverse effects of long-term black raspberry administration of post-surgical HN cancer patients | up to 6 months
  Use diaries and collection of "empties" over 6-month treatment period. Test both measures simultaneously using global test. Two measures tested individually at alpha=0.05 if global test is significant. First check for interaction effect between dose and delivery with double-sided test at alpha=0.01. If that isn't significant, use data from both doses to perform a double-sided alpha=0.05 on difference in compliance between delivery methods. Dose response effect in compliance also tested. Exploring for interaction effects with continued tobacco use vs not and oral cavity patients vs others.
Effects of dose and delivery vehicle on the degree of uptake of black raspberry components in target oral tissues of post-surgical HN cancer patients over time and determine the relationships between adherence/exposure data and uptake. | up to 2 years
  A double-sided test at alpha=0.05 and a mean summary across the repeated measures to test the difference in delivery methods will be used. Relationship between diary compliance and empties records and the two berry components measures over time will be modeled. The critical statistical result from this analysis will be the degree to which the individual patient's trends in the compliance measures correlate with the trends for the two components measured. Interaction effects with continued tobacco use will also be checked.
Correlation between change in gene expression within key regulatory pathways and dose and delivery method | up to 2 years
  Using qRT-PCR measurements for each of 8 genes. Multiple endpoint approach for each gene will be used. Linear mixed models will be used for the repeated measures. Global test at 0.05 to decide superior delivery method. Mean summary statistic across the repeated measures will be used. Interaction effect of dose and delivery tested. Test for interaction of tobacco use at 0.05. Proc Mixed used to estimate both within person (over time changes) and between person relationships across berry components and pathway measures.
Sustainability of the measures within genes found to show significant berry effects beyond the 6-month exposure period | up to 2 years
  Slopes of change (toward baseline) estimated. Hypothesis testing to rule out chance as explanation of changes toward baseline in the berry exposed groups. Relationship between sustainability and the delivery dose studied. Effects on sustainability of continued or changing tobacco use will be estimated. Measures during extended follow-up that are clear indicators of efficacy will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Agrawal, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu